CLINICAL TRIAL: NCT06697379
Title: Key Technology Research and Application Demonstration of Individual Protective Equipment for High-Level Biosafety Laboratories
Status: Active, not recruiting | Type: Observational
Sponsor: Minghui Li (Other Government)
Responsible Party: Sponsor-Investigator, Minghui Li, Doctor, Professor, Beijing Municipal Administration of Hospitals
Organization: Beijing Municipal Administration of Hospitals (Other Government)
Other Study IDs: 2022YFC2603505
Record Dates: First submitted 2024-11-05; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Biosafety Protection; Infectious Diseases
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Systematically evaluate the safety performance, intelligent application effect and experience of PPE developed in different scenarios.

DETAILED DESCRIPTION:
In high-level biosafety laboratories, the National Center for Infectious Disease Medicine, medical consortiums and other national platforms, systematic assessment of the project developed individual physical protection equipment in different scenarios of the safety performance, the intelligent application of the effect and the use of experience, the assessment of the indicators covering the protection performance, safety, stability, comfort, environmental protection, intelligence, ease of operation, including but not limited to local breakage protection performance, Aerosol protection performance, airtightness, liquid penetration performance, differential pressure stability, noise value, air supply flow, ease of wear and removal, ease of movement, ease of operation, degradability, degree of intelligence, etc., and ultimately determine the technical indicators and testing methods of individual physical protective equipment, and establish evaluation technical standards. Based on the determined technical indexes and testing methods of individual physical protective equipment, we will carry out parallel comparative evaluation of similar foreign imported equipment, and form a technical research report on the evaluation of the performance of relevant protective equipment. Optimise the quantitative performance indexes of PPE for domestic shortcomings and weaknesses. Prepare standard operation norms and technical standards for individual physical protective equipment.

ELIGIBILITY:
Inclusion Criteria:

* Staff at outbreak sites, infectious disease wards, BSL-3 and 4 laboratories

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Staff at outbreak sites, infectious disease wards, BSL-3 and 4 laboratories
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Performance evaluation of medical protective clothing | 3 years
  Evaluate the performance of self-developed equipment versus commercially developed equipment, such as protective clothing, hoods, boots and gloves.
  Protective clothing:
  Surface moisture resistance: according to the standard including GB/T 4745-1997 on the level of water, the protective clothing outside the water level is not less than level 3 Hydrostatic pressure: according to GB/T 4744-1997, the hydrostatic pressure is not less than 1.67kPa or 17cmH2O.
  Moisture permeability: according to GB/T 12704-1991, the moisture permeability is not less than 2500g/(m²-24h).
  Water staining test: according to GB/T 4745-1997, the outer water staining level is not less than 3.
  Microbiological barrier performance: the protective clothing should meet the requirements of microbiological indicators in GB 15979-2002 to ensure that it can effectively block the invasion of bacteria, viruses and other microorganisms.

SECONDARY OUTCOMES:
Protective headgear performance evaluation | 3 years
  Protective hood:
  Bacterial filtration efficacy expressed as BFE Rupture strength and elongation at break evaluated in Newtons Moisture permeability is evaluated by m²-24h. Water exposure test: According to GB/T 4745-1997, the external water exposure level should not be less than grade

CONTACTS AND LOCATIONS:
Locations (1):
- Capital medical university, Beijing, Beijing Municipality, China